CLINICAL TRIAL: NCT02334826
Title: Revascularization With the Use of Biodegradable Scaffolds Compared to CABG in Patients With Advanced Stable Ischemic Heart Disease
Brief Title: Revascularization With BVS or CABG in Patients With Advanced CAD
Acronym: RELEASE-BVS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment in one site and withdrawal of the second site prior to enrollment of first participant;
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Maciej Lesiak, MD, PhD, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Poznan01/2015
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Multivessel Coronary Artery Disease
Keywords: multivessel coronary artery disease; revascularization; bioresorbable vascular scaffold; percutaneous coronary intervention; coronary artery bypass grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI - BVS (Active Comparator): percutaneous coronary intervention with the use of bioresorbable scaffolds (Absorb)
  Interventions: Procedure: PCI -BVS
- CABG (Active Comparator): coronary artery bypass grafting
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: PCI -BVS — All patients in the PCI arm will be treated with bioresorbable scaffolds (Absorb). Lesions in native coronary arteries ≥2.25 mm to ≤4.0 mm in diameter (by visual estimate) will be treated after confirmation of functional significance with iFR/FFR.
  Arms: PCI - BVS
Procedure: CABG — In the CABG arm the surgery will be carried out according to the routine practice, with the intention of complete revascularization and frequent use of arterial grafts.
  Arms: CABG

SUMMARY:
The purpose of the study is to investigate the extent of ischemia and left ventricular function in cardiovascular magnetic resonance (CMR), as well as patency of coronary arteries and grafts in coronary computed tomography angiography at 12 months follow up in patients with advanced coronary artery disease treated with percutaneous coronary intervention with the implantation of bioresorbable scaffolds or coronary artery bypass graft surgery.

Additionally, the clinical results of the two methods of revascularization will be carried out annually up to 5 years.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death among adult population in developed countries. Optimal method of revascularization of patients with multivessel CAD is still the matter of debate. Currently, there are two recognized methods: percutaneous coronary intervention (PCI) and coronary artery bypass grafting (CABG). Both methods were compared in a number of studies, including several randomized trials. Most trials have left some doubts. First of all, none of them used functional evaluation of the stenosis. The decision regarding revascularization was based on angiographic results alone. The trials that have used fractional flow reserve (FFR) show no clear correlation between the degree of stenosis assessed angiographically, in the range of 50-90%, and its functional significance. In a randomized FAME trial, out of 1329 significant stenosis assessed anatomically, nearly 40% revealed no functional significance. The study showed that coronary revascularization guided by FFR in multivessel stable CAD resulted in a smaller number of vessels stented, and hence fewer stent implantations. Such a strategy has improved patient clinical outcomes. In the group of patients undergoing revascularization based on fractional flow reserve significant reduction in major adverse cardiac events (MACE) was observed in 1- and 2-year follow up.

Another weakness of former studies was the use of first-generation drug eluting stent (DES) showing an increased risk of restenosis and late and very late stent thrombosis. Many randomized studies documented superiority of new generation DES, with more biocompatible or bioresorbable polymer in terms of the incidence of MACE (SPIRIT, LEADERS). Recently, fully bioresorbable vascular scaffolds (BVS) have been introduced into routine clinical practice. Preliminary results of the ABSORB EXTEND trial demonstrated similar efficacy and safety of the Absorb BVS, as compared with the best-in-class its metallic counterpart XIENCE. Since the complete resorption of the scaffold requires two-three years, the greatest clinical benefit will be observed a couple of years after implantation. Total bioresorption of the scaffold not only allows to restore the physiological function of the vessel, but also eliminates a number of adverse events associated with the presence of permanent metallic prosthesis in the vessel wall, such as very late stent thrombosis and the neo-atherosclerosis development.

Intravascular imaging with intravascular ultrasound (IVUS) or optical coherence tomography (OCT) is widely considered the gold standard for scaffold optimal implantation, although currently it is not routinely used. The use of intravascular imaging techniques before and after BVS implantation may help to avoid inadequate expansion and apposition of the scaffold struts. Subintimal calcifications detected with IVUS or OCT require adequate lesion preparation before stent deployment. This is particularly crucial for patients receiving BVS, where the goal of lesion preparation is to facilitate scaffold delivery, reduce plaque shift and to allow optimal scaffold expansion. OCT with its greater resolution enables to assess the scaffold integrity, apposition and the presence of thrombus or edge dissections.

Based on the ABSORB EXTEND trial there are some suggestions for longer dual antiplatelet therapy duration and more potent agents than clopidogrel (i.e. ticagrelor) regardless of clinical presentation, particularly in the first months after BVS implantation. Ticagrelor in the PLATO trial has been shown to reduce the rate of a combined endpoint of cardio-vascular death, myocardial infarction, or stroke compared to clopidogrel. In patients treated with PCI, it also reduces the rate of stent thrombosis. Statins are the most widely used LDL-lowering drugs in high-risk patients. It is recommended to achieve a greater than 50% reduction in LDL levels. Treatment goal for fasting LDL-cholesterol is < 70 mg/dl (1.8 mmol/l). In comparison with other lipid-lowering agents, rosuvastatin is the most potent agent to achieve the required reduction of LDL. Rosuvastatin in maximal tolerated dose is indicated to reduce the risk of myocardial infarction and revascularization procedures.

RELEASE-BVS study is the first trial that takes into account all of the following important aspects:

* stable advanced coronary artery disease: 3-vessel disease or significant left main (LM) stenosis, suitable for either PCI or CABG with proven ischemia in stress CMR;
* coronary revascularization (PCI) guided by functional assessment of stenosis (iFR/FFR);
* the use of a bioresorbable everolimus-eluting scaffolds (Absorb) and PCI optimization with intracoronary imaging techniques (OCT);
* long-term post-procedural management with potent antiplatelet drug (ticagrelor) and optimal lipid-lowering therapy with maximal tolerated dose of rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 years
* Patient with symptomatic stable CAD or silent ischemia, with 3-vessel disease and/or significant stenosis of left main coronary artery on angiography, with significant ischemia evaluated in stress CMR
* Patient suitable for both PCI or CABG after local heart team evaluation
* Patient understands and accepts the meaning and the aims of the study and is willing to sign written informed consent

Exclusion Criteria:

* Prior CABG
* Concomitant valve disease requiring cardiac surgery
* Metal implants that may be the contraindication for CMR examination (e.g. peacemaker, ICD)
* Other contraindication for stress CMR or computed tomography (claustrophobia, asthma, a-v bloc, allergy to radiographic contrast or any prior anaphylaxis to contrast)
* Contraindication for 12 months dual antiplatelet therapy (DAPT) or known allergy to acetylsalicylic acid, clopidogrel or ticagrelor
* Female patient with child bearing potential
* Acute coronary syndrome within 2 weeks prior to revascularization
* Significant stenosis of any vessel, including LM if reference diameter > 4mm
* left ventricular ejection fraction (LVEF) <35%
* Life expectancy < 12 months
* Stroke or transient ischemic attack (TIA) within 3 months prior to revascularization
* Chronic kidney disease, estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2
* Planned surgery (other than CABG) within 12 months after randomization
* Diathesis, chronic oral anticoagulation therapy or history of bleeding
* Current participation in another trial or registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-02; Primary Completion 2017-09 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Extent of ischemia and left ventricular ejection fraction in cardiovascular magnetic resonance | 12 months after procedure

SECONDARY OUTCOMES:
Patency of coronary arteries and grafts in computed tomography angiography | 12 months after procedure
Rates of composite major adverse cardiac and cerebrovascular events (MACCE), such as all-cause death, cardiac death, myocardial infarction, stroke, stent thrombosis, a repeat revascularization | at 30-day after procedure and annually up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Lesiak, MD, PhD, Principal Investigator — Department of Cardiology, Poznan University of Medical Sciences
Locations (1):
- Department of Cardiology, Poznan University of Medical Sciences, Poznan, Poland